CLINICAL TRIAL: NCT02847949
Title: A Phase 1, Open-Label, Extension Study of Multiple Intravenous Doses of IGN002 Administered Weekly to Subjects With Refractory Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study of IGN002 for Refractory NHL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Reasons
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGN002-201
Record Dates: First submitted 2016-07-12; First posted 2016-07-28 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Extension arm (Experimental): IGN002 study drug will initially be administered at the same dose level and schedule that the subject was receiving at the conclusion of the other Spectrum sponsored IGN002 study, IGN002-101.
  Interventions: Biological: IGN002

INTERVENTIONS:
Biological: IGN002 — IGN002 is a monoclonal antibody fusion protein

SUMMARY:
This is a Phase 1 multi-center, open-label study that allows subjects who derived clinical benefit after completing IGN002 treatment in the Spectrum sponsored IGN002-101 study to continue treatment with IGN002. Subjects who completed the IGN002-101 study, tolerated IGN002 treatment, and did not experience progressive disease (PD) are eligible to participate in this study.

DETAILED DESCRIPTION:
In this extension study, IGN002 study drug will initially be administered at the same dose level and schedule that the subject was receiving at the conclusion of the Spectrum sponsored IGN002-101 study. If additional safety and PK data from another Spectrum sponsored IGN002 study support a higher dose level that is deemed safe and well tolerated by the Safety Review Committee (SRC), the dose of IGN002 may be increased within a given subject. However, dose levels of IGN002 in this extension study may not exceed the maximum tolerated dose (MTD). In addition, the dose for a given subject may be lowered per Investigator discretion. Each treatment cycle comprises a total of 8 doses of IGN002 administered at weekly intervals.

Subjects will be evaluated at the study clinic before each dose of IGN002. At each study visit, standard of care assessments will be performed, which will include physical examination, measurement of vital signs, documentation of adverse events (AEs) and concomitant medications, and laboratory analyses of blood and urine. Radiological assessments will be performed at the end of each 8-week cycle. Tumor status will be assessed by comparison to the subject's baseline tumor status, as determined in the separate study, IGN002-101, or tumor nadir, if the subject has demonstrated response.

Reasons for subject withdrawal include PD in subjects not deriving clinical benefit from IGN002 therapy or clinically significant IGN002-related AEs. If a subject discontinues the study for any reason, an early termination (ET) visit will be conducted 30 (±3) days after the last dose of IGN002. This visit will include physical examination, vital sign measurements, laboratory analyses of blood and urine, and documentation of AEs and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in Spectrum sponsored IGN002 study, IGN002-101
2. Derived clinical benefit from IGN002, defined as CR, PR, or SD, in IGN002-101 study
3. Tolerated IGN002 therapy in the other Spectrum sponsored IGN002 study
4. Female subject is post-menopausal (no menstrual period for a minimum of 12 months) or surgically sterilized and has a negative serum pregnancy test upon entry. Women of childbearing potential (WOCBP) must use an oral or implanted contraceptive, a double barrier method of birth control or an intrauterine device upon enrollment through 3 months after receiving the last dose of IP. Male subject is surgically sterile or is willing to use contraception upon enrollment through 3 months after receiving the last dose of IP.
5. Able and willing to provide informed consent

Exclusion Criteria:

1. Discontinued from other Spectrum sponsored IGN002 study, IGN002-101 due to an AE considered by the Investigator to be related to IGN002 treatment
2. Experienced PD during participation in other Spectrum sponsored study, IGN002-101
3. Pregnant or nursing
4. Concurrent medical condition that precludes safe participation in this study
5. Active viral hepatitis infection. Subjects with history of hepatitis infection that is not active are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence of adverse events following multiple doses of IGN002 administered weekly as an IV infusion to subjects with refractory NHL | An average of 1 year.
  Adverse Event collection and assessment will be done to assess the safety and tolerability of IGN002

SECONDARY OUTCOMES:
Duration of response to IGN002 using the Lugano Classification for NHL | Through study completion, an average of 1 year.
  Lugano Classification Criteria for NHL will be used to assess the duration of response to IGN002
Overall response rate of the therapeutic agent in NHL patients. | Through study completion, an average of 1 year.
  Overall response rate following IGN002 treatment will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: John Timmerman, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No